CLINICAL TRIAL: NCT06961773
Title: Bone Metabolism in Exercising WOMEN: Influence of Low Energy Availability and Sex Hormone Fluctuations
Brief Title: Bone Metabolism in Premenopausal Exercising Women
Acronym: BeWOMEN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, ANA BELEN PEINADO LOZANO, Principal Investigator, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-091
Record Dates: First submitted 2025-03-06; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Contraception; Bone Metabolism; Low Energy Availability; Eumenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eumhenorreic females (Experimental)
  Interventions: Other: Low energy availability; Other: High energy availability
- Oral concetraceptive users (Experimental)
  Interventions: Other: Low energy availability; Other: High energy availability

INTERVENTIONS:
Other: Low energy availability — Participants follow 6 days of a low-energy availability diet. The kilocalories of each diet are prescribed individually based on their fat-free mass.
Other: High energy availability — Participants follow 6 days of a high-energy availability diet. The kilocalories of each diet are prescribed individually based on their fat-free mass.

SUMMARY:
The main goal of this study is to examine how sex hormones and low energy availability affect the concentrations of bone remodelling markers at rest and after a running protocol. The research questions to be addressed are:

1: Does the ovarian hormone profile influence serum bone marker concentrations in women exercising resting and in response to to exercise?

2. Are there differences in response to low energy availability in bone marker concentrations between eumenorrhoeic female athletes and oral contraceptive users?

3: Is the response of bone markers affected by different exercise stimuli: endurance or aerobic endurance?

4: Do bone markers return to baseline levels after 24 hours of high energy availability diet after 6 days of low energy availability?

DETAILED DESCRIPTION:
To achieve the aim of the study, there will be two experimental groups - e.g. eumenorrhoeic females and oral contraceptive users - who, after screening, will be randomly assigned to a low- or high-energy diet. After 6 days on this diet, the participant will undergo an intervallic running protocol and blood samples will be taken before and after the test. The following month the participant will do the other type of diet.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy and between 18 and 30 years old.
* Engage in endurance sports that involve running (such as athletics, running, triathlon, trail running, etc.) for 3 to 12 hours per week..
* Eumenorrheic females with regular menstruation at least 6 months prior to the study.
* Monophasic oral contraceptive users at least 6 months prior to the study.

Exclusion Criteria:

* Amenorrheic females.
* Pregnant females.
* Affected by any disorder related to the hypothalamo-pituitary-ovarian axis.
* Having suffered a bone fracture in the year before the study.
* Taking any medication or supplements that affect bone metabolism.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Concentration of bone metabolism biomarkers | immediately pre-exercise and immediately, 15 minutes and 24 hours post-exercise
  Concentration of procollagen type I N-propeptide (P1NP), cross-linking telopeptide of type I collagen (βCTX-1), paratyroid hormone, calcium, sclerostin, osteoprotegin, osteocalcin, bone alkaline phospatase, Receptor Activator for Nuclear Factor κ B Ligand (RANKL) measured in serum samples.
Concentrations of other biochemical biomarkers | Immediately pre-exercise and immediately, 15 minutes and 24 hours post-exercise
  Concentrations of Triiodothyronine (T3), Albumin, Sex Hormone Binding Globulin (SHBG), etc. measured in serum
Concentrations of sex hormones | Immediately pre-exercise and immediately, 15 minutes and 24 hours post-exercise
  Concentrations of 17β-Oestradiol and Progesterone measured in serum.
Bone mineral density | At the screening phase
  Total, lumbar spine and femoral neck bone mineral density (g/cm^2) measured by dual x-ray absorptiometry

SECONDARY OUTCOMES:
Training status variables | At the screening phase
  Oxygen uptake at ventilatory threshold 1, ventilatory threshold 2, and maximal oxygen uptake (ml/kg/min) measured with a gas analyser.
Body composition variables | Immediately pre- and post-nutritional intervention (bioimpedance) and DXA at the screening
  Fat mass (kg), fat free mass (kg), fat mass percentage, fat-free mass percentage (FFM), total mass (kg) measured by dual x-ray absorptiometry
Body metrics | Measured at the screening phase
  Height (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical activity and sport sciences, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: No